CLINICAL TRIAL: NCT02454829
Title: Follow-up of Ovarian Function in Young Girls and Women Who Underwent Ovarian Cortex Cryopreservation for Fertility Preservation at the Cliniques Universitaires Saint-Luc
Brief Title: Follow-up of Ovarian Function in Young Women Who Underwent Ovarian Cortex Cryopreservation
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: CRYOFONOV01
Record Dates: First submitted 2015-04-22; First posted 2015-05-27 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Female Infertility
Keywords: Ovarian cortex cryopreservation; ovarian function
MeSH Terms: conditions — Infertility, Female | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Adults, gonadotoxic treatment: Women 18 years of age or older who underwent ovarian cortex cryopreservation before gonadotoxic treatment (chemotherapy, radiotherapy)
  Interventions: Other: questionnaire
- Girls, gonadotoxic treatment: Girls under 18 years of age who underwent ovarian cortex cryopreservation before gonadotoxic treatment (chemotherapy, radiotherapy)
  Interventions: Other: questionnaire
- Adults, ovarian pathology: Women 18 years of age or older who underwent ovarian cortex cryopreservation for an ovarian pathology not requiring gonadotoxic treatment but surgery
  Interventions: Other: questionnaire
- Girls, ovarian pathology: Girls under 18 years of age who underwent ovarian cortex cryopreservation for an ovarian pathology not requiring gonadotoxic treatment but surgery
  Interventions: Other: questionnaire
- Adults, genetic disorders: Women 18 years of age or older who underwent ovarian cortex cryopreservation in the context of a genetic risk of premature ovarian failure
  Interventions: Other: questionnaire
- Girls, genetic disorders: Girls under 18 years of age who underwent ovarian cortex cryopreservation in the context of a genetic risk of premature ovarian failure
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — A questionnaire will be send concerning the patient's ovarian function since the cryopreservation procedure i.e: progression of puberty, menstrual cycle, hormonal treatment, desire for pregnancy, occurence of pregnancy, details of pregnancy, need for ART (Artificial Reproductive Techniques), and about the patient's satisfaction concerning the cryopreservation procedure. Data collected will be correlated with treatments received.

SUMMARY:
Evaluation of ovarian function by a questionnaire and by medical file analysis of women and girls who underwent ovarian cortex cryopreservation for fertility preservation between 1997 an 2013 in the investigators' institution in order to evaluate their residual ovarian function. A second part of the questionnaire concerns these women's satisfaction regarding the procedure.

DETAILED DESCRIPTION:
Between 1997 and december 2013, 546 girls and women underwent ovarian cortex cryopreservation in the investigators' institution for fertility preservation. The main indications were the need for a gonadotoxic treatment, repeated ovarian surgery and a genetic risk for premature ovarian failure . These women will be sent a questionnaire concerning their ovarian function since the procedure and a questionnaire about their satisfaction concerning the procedure. Six different questionnaires will be used adapted to the patient's initial indication for cryopreservation and the patient's age at the time of cryopreservation. Complementary data will be obtained by medical file analysis and by contacting the patient's family doctor or gynecologist.

Data will be correlated with received gonadotoxic treatment and surgical interventions.

The purpose of the study is to improve the indications and patient selection for ovarian cortex cryopreservation.

ELIGIBILITY:
Inclusion Criteria:

* women who underwent ovarian cortex cryopreservation in our institution between 1997 and 2013

Exclusion Criteria:

* deceased women in this cohort

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All women who underwent ovarian cortex cryopreservation in our institution between 1997 and 2013
Sampling Method: Non-Probability Sample
Enrollment: 546 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Persistence of ovarian function | since the cryopreservation procedure (24 up to 216 months)
  Prove of ovarian function will be the occurence of pregnancy, the presence of menstrual cycles without hormonal treatment based on the questionnaire or on biological findings compatible with ovarian function in medical file

SECONDARY OUTCOMES:
Satisfaction with the undergone cryopreservation procedure | at the time of completion of the questionnaire (24 up to 216 months after the cryopreservation procedure)
  The questionnaire will evaluate the patient's satisfaction concerning the cryopreservation procedure

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Jadoul, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Belgium